CLINICAL TRIAL: NCT01662102
Title: An Open-Label, Multicenter, Randomized Study in Previously Untreated Follicular Lymphoma Patients to Evaluate the Efficacy of Consolidation With Zevalin® Versus Maintenance Treatment With Rituximab After Initial Therapeutic Response to Rituximab Plus Chemotherapy
Brief Title: Rituximab or Zevalin - Efficacy Trial of Therapeutic Alternatives (RoZetta)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPI-ZEV-12-302
Record Dates: First submitted 2012-08-03; First posted 2012-08-10 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zevalin Regimen Consolidation (Group A) (Experimental): 90Y-Ibritumomab tiuxetan administered 8 to 12 weeks after the last chemotherapy infusion. Each participant randomized to this treatment group was to receive a therapeutic dose of 14.8 MBq/kg (0.4 mCi/kg of total body weight) of 90Y ibritumomab tiuxetan (maximum 1,184 MBq or 32 mCi). Participants with a pre-treatment platelet count between 100 and 149 x10^9/L were to receive 0.3 mCi/Kg 90Y-ibritumomab tiuxetan. (Body weight ≤80 kg: 14.8 MBq [0.4 mCi] yttrium-90/kg and Body weight >80 kg: 1,184 MBq [32 mCi] maximum dose).
  The 90Y ibritumomab tiuxetan regimen is as follows: Day 1 rituximab (250 mg/m^2); Day 7,8, or 9 rituximab (250 mg/m^2) followed by 90Y ibritumomab tiuxetan within 4 hours of the end of the rituximab infusion. (Maximum duration of study was up to approximately 2.7 months).
  Interventions: Drug: Zevalin; Drug: Rituximab
- Rituximab Maintenance (Group B) (Active Comparator): Participants were to receive 375 mg/m^2 of rituximab, administered by intravenous (I.V.) infusion every 8 weeks, starting 8 to 12 weeks after the last R-chemotherapy cycle. (Maximum duration of study was up to approximately 2.7 months).
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Zevalin — Zevalin administered intravenously.
  Other Names: 90Y-ibritumomab tiuxetan
  Arms: Zevalin Regimen Consolidation (Group A)
Drug: Rituximab — Rituximab administered intravenously.
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to evaluate the effect of consolidation treatment Zevalin® versus maintenance treatment with Rituxan® on progression-free survival (PFS) following response induction with chemotherapy plus rituximab in previously untreated participants with follicular lymphoma.

DETAILED DESCRIPTION:
This is an open-label, multicenter and randomized study. Participants registered after response induction (PR/CR) to R-chemotherapy. Participants achieving either a partial response (PR) or complete response (CR) following R-chemotherapy eligible for randomization to either consolidation with 90Y-ibritumumab tiuxetan followed by observation for 24 months, or rituximab maintenance for 24 months. After the observation/maintenance period, patients follow up for 5 years.

This study was terminated early for business reasons. (Maximum duration of study was up to approximately 2.7 months).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age.
* Previously untreated with histologically confirmed grade 1, 2 or 3a cluster of differentiation-20 (CD20)-positive follicular lymphoma, with any of the GELF (Groupe d'Etude de Lymphomes Folliculaires) treatment criteria prior to induction.
* Achieved a response to induction treatment with either rituximab-cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) (6 cycles of R-CHOP21 or R-CHOP14), rituximab-cyclophosphamide, vincristine and prednisone (R-CVP) (6 cycles), or rituximab-bendamustine (R-B) (4 to 6 cycles).
* Must have completed all doses of the induction treatment, except for the modifications allowed in the protocol.

Exclusion Criteria:

* Transformation to high grade lymphoma (secondary to "low grade" follicular lymphoma [FL]).
* Grade 3b follicular lymphoma.
* Primary follicular lymphoma of the skin or gastrointestinal tract.
* Previous treatment of follicular lymphoma.
* Altered renal and hepatic function.
* Known human immunodeficiency virus (HIV) infection and/or active hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection
* Serious co-morbid conditions (for example, ongoing infection, uncontrolled diabetes mellitus, gastric ulcers, active autoimmune disease).
* Life expectancy < 6.
* Must have:

  * Platelet count ≥ 100x10^9/L.
  * Bone marrow infiltration <25%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2013-03-05 (Actual); Study Completion 2013-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cabanillas, MD, Principal Investigator — M.D. Anderson Cancer Center; Thomas Witzig, MD, Principal Investigator — The Mayo Clinic & Foundation; Steven E Finkelstein, MD, Principal Investigator — GenesisCare USA; Leonard Klein, MD, Principal Investigator — Illinois Cancer Specialists - US Oncology; Steven Jubelirer, MD, Principal Investigator — West Virginia University; Petros Nikolinakos, MD, Principal Investigator — Northeast Georgia Cancer Care
Locations (5):
- United States (5):
  - 21st Century Oncology, Sun City, Arizona
  - Northeast Georgia Cancer Care, Athens, Georgia
  - Illinois Cancer Specialists, Niles, Illinois
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Charleston Area Medical Center, Charleston, West Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Zevalin Regimen Consolidation (Group A): 90Y-Ibritumomab tiuxetan administered 8 to 12 weeks after the last chemotherapy infusion. Each participant randomized to this treatment group was to receive a therapeutic dose of 14.8 megabecquerel/kilogram (MBq/kg) (0.4 millicurie/kg [mCi/kg] of total body weight) of 90Y ibritumomab tiuxetan (maximum 1,184 MBq or 32 mCi). Participants with a pre-treatment platelet count between 100 and 149 x10^9/L were to receive 0.3 mCi/Kg 90Y-ibritumomab tiuxetan. (Body weight ≤80 kg: 14.8 MBq [0.4 mCi] yttrium-90/kg and Body weight >80 kg: 1,184 MBq [32 mCi] maximum dose).
  The 90Y ibritumomab tiuxetan regimen is as follows: Day 1 rituximab (250 milligram/meter^2 [mg/m^2]); Day 7,8, or 9 rituximab (250 mg/m^2) followed by 90Y ibritumomab tiuxetan within 4 hours of the end of the rituximab infusion. (Maximum duration of study was up to approximately 2.7 months)
Period: Overall Study
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Sponsor's decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant was enrolled in the Zevalin Regimen Consolidation (Group A) arm. Due to confidentiality considerations, baseline data is not being provided to protect participant privacy.
Groups:
- Zevalin Regimen Consolidation (Group A): 990Y-Ibritumomab tiuxetan administered 8 to 12 weeks after the last chemotherapy infusion. Each participant randomized to this treatment group was to receive a therapeutic dose of 14.8 MBq/kg (0.4 mCi/kg of total body weight) of 90Y ibritumomab tiuxetan (maximum 1,184 MBq or 32 mCi). Participants with a pre-treatment platelet count between 100 and 149 x10^9/L were to receive 0.3 mCi/Kg 90Y-ibritumomab tiuxetan. (Body weight ≤80 kg: 14.8 MBq [0.4 mCi] yttrium-90/kg and Body weight >80 kg: 1,184 MBq [32 mCi] maximum dose).
  The 90Y ibritumomab tiuxetan regimen is as follows: Day 1 rituximab (250 mg/m^2); Day 7,8, or 9 rituximab (250 mg/m^2) followed by 90Y ibritumomab tiuxetan within 4 hours of the end of the rituximab infusion. (Maximum duration of study was up to approximately 2.7 months)
- Total: Total of all reporting groups
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) is defined as the time from randomization until progression, relapse, death from any cause, or introduction of a new anti-lymphoma treatment (chemotherapy, radiation therapy or immunotherapy).
Time Frame: Up to approximately 2.7 months
Population: Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Complete Response Rate
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Event Free Survival
Description: EFS time is defined as the time from randomization to first documented progression, death from any cause, or introduction of a new anti-lymphoma treatment (chemotherapy, radiotherapy or immunotherapy).
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from randomization to the first disease progression.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Next Anti-Lymphoma Treatment (TTNLT)
Description: TTNLT is defined as the time from randomization to the first introduction of any new anti lymphoma regimen.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Next Chemotherapy (TTNCT)
Description: TTNCT is defined as the time from randomization to the first introduction of any new chemotherapy (cytotoxic or radioimmunotherapy). The TTNCT may be the same as the TTNLT. Participants who respond to treatment and Participants who are lost to follow-up censored at the visit on which the dosing of a new medication was evaluated.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Response Rate (ORR)
Description: Tumor response evaluated according to Cheson criteria at the time of randomization and at the end of the maintenance/observation, post randomization. ORR is defined as the percentage of Participants with a complete response (CR) or a partial response (PR), and compared between treatment groups. Participants with no response evaluation (for any reason) considered as not evaluable (NE).
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause. In living patients, survival time was censored on the last date participants were known to be alive.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Transformation at First Progression
Description: Transformation rate at first progression, defined as the appearance of diffuse areas of large lymphoma cells within a tumor site.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Toxicity
Description: Toxicity graded according to the National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.0.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With Secondary Malignancies
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Functional Assessment of Cancer - General (FACT-G)
Description: The FACT-G is a participant rated, 27-item compilation of general questions divided into 4 primary Quality of Life (QOL) sub-scales: physical well-being (PWB; 7-items, score range 0-28), social/family well-being (SWB; 7-items, score range 0-28), emotional well-being (EWB; 6-items, score range 0-24), and functional well-being (FWB; 7-items, score range 0-28). This tool represents the generic core questionnaire that are utilized in combination with cancer site-specific questionnaires, (FBrain, in this study) Overall score and four subscale scores with ranges and distributions that are sample-specific can be calculated.FACT-G is scored by summing the individual scale scores; higher scores indicate better quality of life. FACT-G uses 5-point rating scale ranging from (0) = Not at all; (1) = A little bit; (2) = Somewhat; (3) = Quite a bit; to (4) = Very much.The FACT-G total score is the sum of the four subscale scores (if least 80% completed) and has a possible range of 0-108 points.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC-QLQ-C30 is a cancer-specific instrument with 30 questions for evaluation of new chemotherapy and provides an assessment of participant reported outcome dimensions. First 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical,role,emotional,cognitive,social), 3 symptom scales (fatigue,nausea/vomiting,pain) & other single items. For each item,high score represented high level of symptomatology/problem. Last 2 questions represented participant's assessment of overall health & quality of life, coded on 7-point scale (1=very poor to 7=excellent).EORTC QLQ-C30 observed values and change from baseline for global health status (scoring of questions 29 & 30) and 5 functional scales, 3 symptom scales and other single items (scoring of questions 1 to 28). Answers were converted into grading scale, with values between 0 and 100. High score represented a favourable outcome with a best quality of life for participant.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Pharmacoeconomics (Cost Effectiveness Analysis)
Description: A cost-effectiveness analysis done that compares the efficiency (cost/effectiveness unit) of consolidation treatment with 90Y-ibritumomab tiuxetan compared to maintenance treatment with rituximab. The analysis conducted according to a health economic analysis plan independent from this clinical study protocol.
Time Frame: Up to approximately 2.7 months
Population: as for outcome 1
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 2.7 months
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Due to the low number of participants enrolled at only 1 site, 0 participants are reported due to the risk of identification of a person.
Arm/Group | Zevalin Regimen Consolidation (Group A) | Rituximab Maintenance (Group B)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No